CLINICAL TRIAL: NCT04445285
Title: Double Blind Randomized Phase 2 Placebo Controlled Trial Using rhDNase to Reduce Mortality in COVID-19 Patients With Respiratory Failure
Brief Title: Phase 2 Trial Using rhDNase to Reduce Mortality in COVID-19 Patients With Respiratory Failure
Acronym: DAMPENCOVID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jon Simmons (Other)
Collaborators: University of South Alabama (Other)
Responsible Party: Sponsor-Investigator, Jon Simmons, Chief, Division of Trauma & Acute Care Surgery, University of South Alabama
Organization: University of South Alabama (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USAH 1002 000
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Covid-19, Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — dornase alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Patient will receive 2.5mg Pulmozyme/ Recombinant human deoxyribonuclease (rh-DNase) aerosolized treatment once every 24 hours for five (5) consecutive days; a total of five (5) doses.
  Interventions: Drug: Pulmozyme/ Recombinant human deoxyribonuclease (rh-DNase)
- Placebo Arm 0.9% sodium chloride (Placebo Comparator): Patient will receive 2.5ml of Sodium Chloride 0.9% aerosolized treatment once every 24 hours for five (5) consecutive days; a total of five (5) doses.
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: Pulmozyme/ Recombinant human deoxyribonuclease (rh-DNase) — 2.5mg Pulmozyme/ Recombinant human deoxyribonuclease (rh-DNase) aerosolized treatment once every 24 hours for five (5) consecutive days; a total of five (5) doses
  Arms: Treatment Arm
Drug: 0.9%sodium chloride — Placebo of 0.9% sodium chloride every 24 hours for five (5) consecutive days; a total of 5 doses
  Arms: Placebo Arm 0.9% sodium chloride

SUMMARY:
This Phase 2 Randomized Placebo Controlled Trial will determine if administering nebulized Dornase Alpha (rhDNase) to COVID-19 patients with respiratory failure is safe and will reduce 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 18 or older
2. On high flow oxygen =/> 6 liters nasal cannula (or)
3. On mechanical ventilation
4. Clinical diagnosis of COVID-19 & positive PCR test (or)
5. Clinical diagnosis of COVID-19 & negative PCR test with clinical symptoms of COVID-19 and pathognomonic lesions on a chest CT scan

Exclusion Criteria:

1. Known allergy to Pulmozyme
2. Less than 18 years of age
3. Grave condition with anticipated death within 48 hours; at the discretion of treating physician.
4. Enrollment in another clinical trial receiving investigatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality at 28 days | 28 days after enrollment
  All Cause Mortality at 28 days
Systemic Therapeutic Response | 5 days after enrollment
  To assess the effect of Pulmozyme® on the severity of respiratory failure, systemic inflammatory response, and multi-organ failure.

SECONDARY OUTCOMES:
Respiratory Response | 28 days
  Proportion of patients alive and free of invasive mechanical ventilation at 28 days invasive mechanical ventilation at 28 days
Legnth of ICU Stay | 28 days
  Proportion of patients alive and discharged from the ICU at 28 days discharged from the ICU at 28 days
Legnth of Hospital Stay | 28 days
  Proportion of patients alive and discharged from the hospital at 28 days
Respiratory Response | 28 days
  Alive, respiratory failure-free days at 28 days
Pulmonary Function | 5 days
  Pulmonary Function Ratio at 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simmons JD, Lee YL, Mulekar S, Kuck JL, Brevard SB, Gonzalez RP, Gillespie MN, Richards WO. Elevated levels of plasma mitochondrial DNA DAMPs are linked to clinical outcome in severely injured human subjects. Ann Surg. 2013 Oct;258(4):591-6; discussion 596-8. doi: 10.1097/SLA.0b013e3182a4ea46. PMID 23979273
- [Background] Zhang Q, Raoof M, Chen Y, Sumi Y, Sursal T, Junger W, Brohi K, Itagaki K, Hauser CJ. Circulating mitochondrial DAMPs cause inflammatory responses to injury. Nature. 2010 Mar 4;464(7285):104-7. doi: 10.1038/nature08780. PMID 20203610
- [Background] Schumacker PT, Gillespie MN, Nakahira K, Choi AM, Crouser ED, Piantadosi CA, Bhattacharya J. Mitochondria in lung biology and pathology: more than just a powerhouse. Am J Physiol Lung Cell Mol Physiol. 2014 Jun 1;306(11):L962-74. doi: 10.1152/ajplung.00073.2014. Epub 2014 Apr 18. PMID 24748601
- [Background] Kuck JL, Obiako BO, Gorodnya OM, Pastukh VM, Kua J, Simmons JD, Gillespie MN. Mitochondrial DNA damage-associated molecular patterns mediate a feed-forward cycle of bacteria-induced vascular injury in perfused rat lungs. Am J Physiol Lung Cell Mol Physiol. 2015 May 15;308(10):L1078-85. doi: 10.1152/ajplung.00015.2015. Epub 2015 Mar 20. PMID 25795724
- [Background] Dobson AW, Grishko V, LeDoux SP, Kelley MR, Wilson GL, Gillespie MN. Enhanced mtDNA repair capacity protects pulmonary artery endothelial cells from oxidant-mediated death. Am J Physiol Lung Cell Mol Physiol. 2002 Jul;283(1):L205-10. doi: 10.1152/ajplung.00443.2001. PMID 12060578
- [Background] Ruchko MV, Gorodnya OM, Zuleta A, Pastukh VM, Gillespie MN. The DNA glycosylase Ogg1 defends against oxidant-induced mtDNA damage and apoptosis in pulmonary artery endothelial cells. Free Radic Biol Med. 2011 May 1;50(9):1107-13. doi: 10.1016/j.freeradbiomed.2010.10.692. Epub 2010 Oct 20. PMID 20969951
- [Background] Chouteau JM, Obiako B, Gorodnya OM, Pastukh VM, Ruchko MV, Wright AJ, Wilson GL, Gillespie MN. Mitochondrial DNA integrity may be a determinant of endothelial barrier properties in oxidant-challenged rat lungs. Am J Physiol Lung Cell Mol Physiol. 2011 Dec;301(6):L892-8. doi: 10.1152/ajplung.00210.2011. Epub 2011 Sep 2. PMID 21890512
- [Background] Gebb SA, Decoux A, Waggoner A, Wilson GL, Gillespie MN. Mitochondrial DNA damage mediates hyperoxic dysmorphogenesis in rat fetal lung explants. Neonatology. 2013;103(2):91-7. doi: 10.1159/000342632. Epub 2012 Nov 15. PMID 23154780
- [Background] Hashizume M, Mouner M, Chouteau JM, Gorodnya OM, Ruchko MV, Potter BJ, Wilson GL, Gillespie MN, Parker JC. Mitochondrial-targeted DNA repair enzyme 8-oxoguanine DNA glycosylase 1 protects against ventilator-induced lung injury in intact mice. Am J Physiol Lung Cell Mol Physiol. 2013 Feb 15;304(4):L287-97. doi: 10.1152/ajplung.00071.2012. Epub 2012 Dec 14. PMID 23241530
- [Background] Simmons JD, Freno DR, Muscat CA, Obiako B, Lee YL, Pastukh VM, Brevard SB, Gillespie MN. Mitochondrial DNA damage associated molecular patterns in ventilator-associated pneumonia: Prevention and reversal by intratracheal DNase I. J Trauma Acute Care Surg. 2017 Jan;82(1):120-125. doi: 10.1097/TA.0000000000001269. PMID 27787436
- [Background] Grishko V, Solomon M, Wilson GL, LeDoux SP, Gillespie MN. Oxygen radical-induced mitochondrial DNA damage and repair in pulmonary vascular endothelial cell phenotypes. Am J Physiol Lung Cell Mol Physiol. 2001 Jun;280(6):L1300-8. doi: 10.1152/ajplung.2001.280.6.L1300. PMID 11350811